CLINICAL TRIAL: NCT01603303
Title: Preventing Sexual Dysfunction in Women on Aromatase Inhibitors
Brief Title: Preventing Sexual Dysfunction With Aromatase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Fidia Farmaceutici s.p.a. (Industry); Laclede, Inc. (Industry); Duncan Family Institute Seed Money Grant (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0125; NCI-2014-02451 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-05-17; First posted 2012-05-22 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Localized breast cancer; Postmenopausal women; Aromatase inhibitor; AI; Questionnaires; Surveys; Luvena; Internet based website; Phone counseling; Water-based vaginal lubricant; Hyalo-Gyn
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care + Education Materials (Other): Completion of 8 or 9 brief questionnaires at start of study and 6 and 12 months afterwards. Questionnaires should take about 45 to 50 minutes to fill out each time. Participants receive written handout about ways to keep bones stronger during treatment with Aromatase Inhibitors (AIs) and ways to prevent AI side effects such as muscle aches, stiffness, sexual problems, and hot flashes. Water-based vaginal lubricant used during sexual activity.
  Interventions: Behavioral: Questionnaires; Other: Education Materials
- Luvena Group (Experimental): Luvena used vaginally 2 or 3 times a week. Completion of 8 or 9 brief questionnaires at start of study and 6 and 12 months afterwards. Questionnaires should take about 45 to 50 minutes to fill out each time. Participants receive written handout about ways to keep bones stronger during treatment with Aromatase Inhibitors (AIs) and ways to prevent AI side effects such as muscle aches, stiffness, sexual problems, and hot flashes. Participants use an interactive, internet-based website called Tendrils: Sexual Renewal after Cancer before, during and after treatment with AIs. Telephone counseling for up to 30 minutes in weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24. The counselor will follow a manualized program and some sessions will be recorded.
  Interventions: Behavioral: Questionnaires; Other: Education Materials; Other: Luvena; Other: Vaginal Lubricant; Behavioral: Interactive Internet-Based Website; Behavioral: Telephone Counseling.
- Hyalo-Gyn Group (Experimental): Hyalo-Gyn used vaginally 2 - 3 times a week. Completion of 8 or 9 brief questionnaires at start of study and 6 and 12 months afterwards. Questionnaires should take about 45 to 50 minutes to fill out each time. Participants receive written handout about ways to keep bones stronger during treatment with Aromatase Inhibitors (AIs) and ways to prevent AI side effects such as muscle aches, stiffness, sexual problems, and hot flashes. Participants use an interactive, internet-based website called Tendrils: Sexual Renewal after Cancer before, during and after treatment with AIs. Telephone counseling for up to 30 minutes in weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24. The counselor will follow a manualized program and some sessions will be recorded.
  Interventions: Behavioral: Questionnaires; Other: Education Materials; Other: Hyalo-Gyn; Other: Vaginal Lubricant; Behavioral: Interactive Internet-Based Website; Behavioral: Telephone Counseling.

INTERVENTIONS:
Behavioral: Questionnaires — Completion of 8 or 9 brief questionnaires at start of study and 6 and 12 months afterwards. Questionnaires should take about 45 to 50 minutes to fill out each time.
  Other Names: Surveys
Other: Education Materials — Participants receive written handout about ways to keep bones stronger during treatment with Aromatase Inhibitors (AIs) and ways to prevent AI side effects such as muscle aches, stiffness, sexual problems, and hot flashes.
  Other Names: Pamphlets
Other: Luvena — Use vaginally 2 or 3 times a week.
  Arms: Luvena Group
Other: Hyalo-Gyn — Use vaginally 2 - 3 times a week.
  Arms: Hyalo-Gyn Group
Other: Vaginal Lubricant — Water-based vaginal lubricant used during sexual activity.
  Arms: Hyalo-Gyn Group; Luvena Group
Behavioral: Interactive Internet-Based Website — Participants use an interactive, internet-based website called Tendrils: Sexual Renewal after Cancer before, during and after treatment with AIs.
  Arms: Hyalo-Gyn Group; Luvena Group
Behavioral: Telephone Counseling. — Telephone counseling for up to 30 minutes in weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24. The counselor will follow a manualized program and some sessions will be recorded.
  Arms: Hyalo-Gyn Group; Luvena Group

SUMMARY:
Aromatase inhibitors (AIs) are used to try to stop breast cancer from forming or returning after treatment in women who are in menopause and who had breast cancer that was sensitive to the hormone estrogen.

The goal of this study is to learn if it is possible to prevent some AI side effects, particularly problems with vaginal dryness and pain during sexual activity. Researchers also want to compare 2 new vaginal moisturizers to see if using them regularly helps women avoid vaginal dryness. Researchers want to see if preventing these side effects will decrease the number of women who stop taking AIs due to the side effects they cause.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be randomly assigned (as in a roll of dice) to 1 of 2 study groups. You will have a 1 in 3 chance of being assigned to Group 1 and a 2 out of 3 chance of being assigned to Group 2.

All women enrolled in this study:

* You will complete a set of 8 or 9 brief questionnaires at the start of the study and 6 and 12 months afterwards. The questionnaires should take about 45 to 50 minutes to fill out each time. The questionnaires will be mailed to you with a postage paid return envelope. They include questions about your background and medical history, any symptoms that you may have while taking AIs such as hot flashes, muscle pain, and stiffness. There are also questions about how much exercise you are getting, sexual function and satisfaction, your satisfaction with the treatment you are receiving as part of this study, and if you are continuing to take your AI medication and how often you are taking it. If the study staff does not receive your questionnaires within 2 weeks of mailing them, you will receive reminder phone calls once a week for up to 3 weeks unless you tell the study staff that you are leaving the study. If you do not contact the study staff or you do not mail in your questionnaires after 6 weeks, you will no longer be a part of the study.
* Along with your questionnaires, you will also be mailed a kit approved by the Food and Drug Administration (FDA) to test your vaginal pH at home and will be provided a postage paid return envelope to mail it back to the study doctor. The kit includes a small plastic stick that you put into your vagina for a moment to test your vaginal fluid. The end of the stick turns different colors, depending on the pH in your vagina. The vagina becomes less acidic after menopause, which may increase the risk of vaginal infections. Sometimes vaginal moisturizers can correct this problem by restoring a pH similar to what it was before menopause.
* You will also receive a detailed written handout about ways to keep your bones stronger during treatment with AIs and ways to prevent AI side effects such as muscle aches, stiffness, sexual problems, and hot flashes.

Group 2 women only:

* You will be given a password to use an interactive, internet-based website called Tendrils: Sexual Renewal after Cancer (https://www.tendrilssexandcancer.com/) before, during and after treatment with AIs. You will also be given a printed guide for the website with a timeline for when you should read certain sections and suggestions for trying some of the "exercises" to improve sexual communication, increase affection, and prevent vaginal dryness.
* A counselor will also schedule times to call you for up to 30 minutes during Weeks 2, 4, 6, 8, 10, 12, 16, 20, and 24 of the study to ask how you are doing, if you have been able to avoid side effects from the AIs, and if you need any help using the information in your handout or the website. About 1 of 5 counseling phone calls will be audio-recorded so that researchers can make sure the counselor is covering the topics scheduled for each session. These recordings will usually only be heard by the counselor, the Study Chair, and another MD Anderson faculty member (Andrea Bradford, PhD) who will help with supervising and rating the counselor. Once a tape has been rated (usually within one month of the counseling session), it will be erased. The tape may also be reviewed by other health authorities or the Institutional Review Board (IRB) of MD Anderson to check that the research is being done safely and correctly. If either of these 2 groups review the tapes, the will be destroyed right after they are reviewed. Tapes will only be labelled by your study number, but the counselor may call you by name during the session. All information will be held in strict confidentiality by research staff.
* You will be randomly assigned (as in the toss of a coin) to get a 6-month supply of 1 of 2 vaginal moisturizers (Luvena or Hyalo-Gyn) to use 2 or 3 times a week. Researchers want to know if one works better than the other for women on AIs.
* You will be given a 6-month supply of a water-based vaginal lubricant to use during sexual activity.
* You will also be given a vaginal dilator, which is used to help women to relax their pelvic floor muscles and to increase blood flow into the vaginal walls.
* All of the materials that you need for the study, including handouts, instructions on using the web site, instructions on using the vaginal moisturizer, vaginal lubricant, and vaginal dilator, as well as the supply of those products, will be mailed to you in a study kit as soon as you complete your baseline questionnaires.

All of your questionnaires and other study records will be identified only with a study number and will not include your name, address, or MD Anderson patient number. A list linking your study number to your identity will be kept either in a locked file cabinet or encrypted on a secure computer. Only the study chair and research staff will be able to see the list. Once all data has been analyzed (May 2015 is the estimated date of completion), these lists will be destroyed. Questionnaires or computer files that identify data only by study number may be kept for up to 10 years to satisfy government rules for research.

Length of Study:

Your active study participation will be over after you complete the questionnaires at 12 months.

Other Information:

You are not required to use the vaginal dilator, the moisturizer, or the lubricant in order to take part in this study, but you will be asked if these products were helpful to you.

This is an investigational study.

Up to 168 women will take part in this study. All will be enrolled at MD Anderson Cancer Center or at MD Anderson Cooper Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Stage 0 to III breast cancer
2. Age over 18 years
3. Began adjuvant therapy with an aromatase inhibitor 12 to 18 months before survey sent out (Benchmark Survey only)
4. Was prescribed adjuvant therapy with an AI (prior chemotherapy or tamoxifen OK) in past 2 to 4 weeks (Randomized Trial only)
5. Had sexual activity at least once in past 12 months (Randomized Trial Study only)
6. Has been in a stable sexual relationship of at least 6 months' duration (Randomized Trial study only)

Exclusion Criteria:

1. Women using systemic or vaginal estrogen, testosterone, or dehydroepiandrosterone (DHEA) during the Randomized Trial study will be excluded
2. Women using systemic or vaginal estrogen, testosterone, or dehydroepiandrosterone (DHEA) in the 12 months preceding the Benchmark Survey Study will be excluded
3. Has distant metastases
4. Cannot read or speak English well enough to understand materials and complete questionnaires
5. No access to the internet in a private location

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2012-12-05 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Sexual Dysfunction Rate Reduction | 12 months
  The primary outcome measure will be the total score from the Female Sexual Function Index (FSFI), which is calculated according to a standard scoring algorithm and has a well-validated cut-off score of 26.55 or below indicating sexual dysfunction. FSFI subscale scores will also be calculated and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Abenaa M. Brewster, MD, MHS, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org